

## Clinical Development

## PKC412/Midostaurin/Rydapt®

CPKC412A2408 / NCT03379727

An open-labeled, multi-center, Phase IIIb study to assess the safety and efficacy of midostaurin (PKC412) in patients 18 years of age or older with newly-diagnosed FLT3-mutated Acute Myeloid Leukemia who are eligible for "7+3" or "5+2" chemotherapy

Statistical Analysis Plan (SAP) – Amendment 3

Author: (Trial Statistician)

Document type: SAP Documentation

Document status: V4.0

Release date: 09-Nov-2021

Number of pages: 30

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

## **Document History – Changes compared to previous final version of SAP**

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 22-Aug-2017 | Prior to<br>FPFV | N/A – Initial version | N/A | N/A |
| 14-Jan-2020 | Prior to<br>database<br>lock | Rules to select one<br>assessment among<br>several assessments in<br>the same visit<br>Time windows for | Selection of assessment to<br>analyze among multiple<br>values in the same visit Time windows to assign | 2.1.5 |
| | | unplanned visits | unplanned visits in scheduled ones | |
| | | Added rules to assign patients to 7+3 and 5+2 groups | Patients who do not have exactly 7+3 or 5+2 are assigned | 2.1.8 |
| | | Category/Value missing | Added treatment exposure category ">28".Cardiac imaging changed ">" to ">-" for 20 | 2.4.2<br>2.8.4.2 |
| | | Change in CSR template | Concomitant medications will be analyzed with FAS instead of SAF | 2.4.3 |
| | | Clinical efficacy<br>response derivation and<br>subgroup analyses | Selection of best response<br>among several assessment<br>in the same period.<br>Response analyzed by sex | 2.6.1 |
| | | AEs by subgroup | AEs to be analyzed by age category | 2.8.1 |
| | | Resource utilization updated to CRF | Updated with variables only included in CRF | 2.13.3 |
| | | Additional details on imputation rules | Derivation rules updated | 6.1 |
| | | BUN/Urea imputation rules | To impute BUN or Urea missing values | 6.2 |
| 26-Jun-2020 | | Study treatment exposure | Rules od study treatment exposure clarified. | 2.1.1 |
| | | Analysis set | All enrolled subjects added | 2.2 |
| | | Subgroups analyses added: type of induction drugs | Efficacy and safety outputs provided by Idarubicin and Daunorubicin. | 2.3 |
| | | Age subgroups | <= 60 vs. >60 instead of <60 vs. >=60 | 2.3 and 2.4.2 |

| Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|
| | Efficay | If patient discontinued prior<br>to first efficacy assessment<br>then 'unknown' is assigned<br>as best response | 2.7.1 |
| = | | | |
| Prior to<br>database<br>lock | PD | The number (%) of protocol deviations with COVID-19 relationship will be presented by type of deviation for all enrolled subjects. | 2.5.4 |
| Post to<br>database<br>lock | Subgroups analysis amended for a new agesubgroup/category. | Included the following age subgroup/category: | 2.3, 2.4.2, 2.5.2 and 2.7.1 |
| | | <= 60 / > 60 to <= 70 / > 70 years old | |
| | Prior to database lock Post to database | Prior to database lock Post to database amended for a new | Prior to database lock Post to Subgroups analysis amended for a new lock Subgroup/category. Efficay If patient discontinued prior to first efficacy assessment then 'unknown' is assigned as best response The number (%) of protocol deviations with COVID-19 relationship will be presented by type of deviation for all enrolled subjects. Included the following age subgroup/category: <= 60 / >60 to <=70 / > 70 |

## **Table of contents**

| 1 | Introd | luction | | 7 |
|---|---|---|---|---|
| | 1.1 | Study o | lesign | 7 |
| | 1.2 Study objectives and endpoints | | objectives and endpoints | 9 |
| 2 | Statis | tical metl | hods | 9 |
| | 2.1 | Data ar | nalysis general information | 9 |
| | | 2.1.1 | General definitions | 9 |
| | | 2.1.2 | Baseline | 13 |
| | | 2.1.3 | On-treatment assessment/event | 13 |
| | | 2.1.4 | Definition of months and years | 14 |
| | | 2.1.5 | Time windows | 14 |
| | | 2.1.6 | Definition of end of study | 15 |
| | | 2.1.7 | Early study termination | 15 |
| | | 2.1.8 | Chemotherapy group assignment | 15 |
| | 2.2 | Analys | is sets | 15 |
| | | 2.2.1 | All enrolled patients | 15 |
| | | 2.2.2 | Full analysis set | 15 |
| | | 2.2.3 | Safety set | 15 |
| | 2.3 | Subgro | oup analysis | 16 |
| | 2.4 | Patient | disposition, demographics and other baseline characteristics | 16 |
| | | 2.4.1 | Patient disposition | 16 |
| | | 2.4.2 | Patient demographics and other baseline characteristics | 16 |
| | 2.5 | Treatm | ents (study treatment, concomitant therapies, compliance) | 16 |
| | | 2.5.1 | Dosing regimen | 16 |
| | | 2.5.2 | Study treatment and tolerability | 17 |
| | | 2.5.3 | Prior, concomitant and post therapies | 18 |
| | | 2.5.4 | Protocol deviations | 18 |
| | 2.6 | Analys | is of the primary objective | 18 |
| | | 2.6.1 | Primary endpoint | 18 |
| | | 2.6.2 | Statistical hypothesis, model, and method of analysis | 18 |
| | | 2.6.3 | Handling of missing values/censoring/discontinuations | 18 |
| | | 2.6.4 | Supportive analyses | 18 |
| | 2.7 | Analys | is of the secondary objectives | 19 |
| | | 2.7.1 | Secondary endpoints | 19 |
| | | 2.7.2 | Statistical hypothesis, model, and method of analysis | 19 |
| | | 2.7.3 | Handling of missing values/censoring/discontinuations | 19 |

| | 2.8 | Analysi | is of secondary efficacy objective(s) | 19 |
|---|-------|------------|---------------------------------------|----|
| | 2.9 | Safety a | analyses | 19 |
| | | 2.9.1 | Adverse events (AEs) | 19 |
| | | 2.9.2 | Deaths | 21 |
| | | 2.9.3 | Laboratory data | 21 |
| | | 2.9.4 | Other safety data | 22 |
| | 2.10 | Pharma | acokinetic endpoints | 23 |
| | 2.11 | PD and | l PK/PD analyses | 24 |
| | | | | 24 |
| | 2.13 | Biomar | rkers | 24 |
| | 2.14 | Other E | Exploratory analyses | 24 |
| | | | | 24 |
| | | | | 25 |
| | | 2.14.3 | Resource utilization | 25 |
| | 2.15 | Interim | analysis | 25 |
| 3 | Samp | le size ca | llculation | 25 |
| 4 | Chang | ge to prot | tocol specified analyses | 26 |
| 5 | Refer | ences | | 26 |
| 6 | Apper | ndix | | 27 |
| | 6.1 | Imputat | tion rules | 27 |
| | | 6.1.1 | AE, CM date imputation | 27 |
| | | 6.1.2 | Prior therapies date imputation | 28 |
| | 6.2 | Laborat | tory parameters derivations | |
| | | | | 28 |

#### List of abbreviations

AE adverse event

AESI adverse events of special interest

ALT aspartate aminotransferase AML acute myeloid leukemia

Ara-C cytarabine, also known as cytosine arabinoside

AST alanine aminotransferase

ATC anatomical therapeutic chemical classification

CIVI continuous intravenous infusion

CR complete remission

CRi complete remission with incomplete recovery

CRS case retrieval sheet CSR clinical study report

CTCAE common terminology criteria for adverse events

DI dose intensity
ECG electrocardiogram

ECOG eastern cooperative oncology group

eCRF electronic case report form

FAS full analysis set

FLT3 fms-like tyrosine kinase receptor

GPS global programming & statistical environment

IV intravenous

LPLV last patient last visit

LVEF left ventricular ejection fraction

MedDRA medical dictionary for drug regulatory affairs

MUGA multi gated acquisition scan

NCCN national comprehensive cancer network

NCDS Novartis clinical data standards

PD pharmacodynamics

PDS programming data specifications

PK pharmacokinetics

PT preferred term

QTc corrected QT interval
SAE serious adverse event
SAP statistical analysis plan
SI international system of units

SOC system organ class
TFLs tables, figures, listings
WHO world health organization

## 1 Introduction

This statistical analysis plan (SAP) provides detailed statistical methodology for the analyses of data which will be used for preparation of the PKC412A2408 clinical study report (CSR) and is based on the study protocol Amendment 1, dated 26-Mar-2018. At the time of this amendment, enrollement was completed with 301 patients.

The shells for the in-text tables and figures as well as the post-text tables, figures and listings (TFLs) are in the TFL shells document. Programming specifications for datasets, including derivation of variables, are given in the programming data specifications (PDS) document.

All data will be analyzed by Novartis using Novartis clinical data standards (NCDS). Analysis data sets and statistical outputs will be produced using the SAS system Version 9.4 or higher (UNIX environment) in the global programming & statistical (GPS) environment.

## 1.1 Study design

This is an open-label, single arm, multicenter, Phase IIIb study of midostaurin (PKC412 or CGP41251) in adults with newly-diagnosed fms-like tyrosine kinase receptor (FLT3)-mutated acute myeloid leukemia (AML) who have started on "7+3" or "5+2" induction chemotherapy.

The purpose of this study is to gather and evaluate additional safety and efficacy data on the combination of midostaurin and standard of care.

Midostaurin is used in combination with chemotherapy sequentially in **induction** and **consolidation** phase and as a single agent in **maintenance** phase as outlined in Figure 1-1.

Approximately 300 patients are planned to be enrolled.

No formal interim analyses are planned.

The final (primary) analysis will be performed after database lock when all patients have either completed the study as per protocol (including their safety evaluation 30 days after the last dose of study treatment) or they have prematurely discontinued.

Figure 1-1 Study design



Complete remission (CR): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) >1.0 x10 $^{9}$ /L; platelet count >100 x 10 $^{9}$ /L; independence of red cell transfusions

CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia (<1.0  $\times$ 10 $^{9}$ /L) or thrombocytopenia (<100  $\times$  10 $^{9}$ /L)

Figure 1-2 Recovery periods



| Objective | Endpoint |
|---|---|
| Primary | |
| To further assess the safety of midostaurin in induction, consolidation and maintenance therapy, including, the "7+3" regimen, daunorubicin (60-90mg/m²/day), the substitution of daunorubicin by idarubicin (12mg/m²/day), cytarabine (100-200 mg/m²/day) and also allowing the "5+2" reduced dose regimen. | Proportion of patients with AEs, Grade 3&4 AEs, SAEs, AEs leading to discontinuation, and deaths. |
| Secondary | |
| To assess the clinical efficacy of midostaurin in combination with chemotherapy regimens in induction and consolidation and the clinical efficacy of midostaurin maintenance phase (measured by CR/CRi rate). | Proportion of patients with CR/CRi as per local assessment |
| Exploratory | |
| To assess resource utilization | Proportion of patients by reason for hospitalization, number of hospital days, discharge reason and concomitant medications taken during hospital stay |
| AE: adverse event | |

## 2 Statistical methods

## 2.1 Data analysis general information

Categorical data will be presented as frequencies and percentages. For continuous data, n, mean, standard deviation, median, 25th and 75th percentiles, minimum, and maximum will be presented.

The data from all centers that participate will be combined in the analyses.

Final (primary) analysis will be performed after database lock has occurred (after last patient last visit (LPLV)).

## 2.1.1 General definitions

The overall observation period is divided into the following mutually exclusive periods:

1. **Pre-treatment**: from day of patient's informed consent to the day before first dose of midostaurin

2. **On-treatment**: from start date of midostaurin to last date of study treatment + 30 days. Further details provided in Section 2.1.3.

On-treatment includes 3 mutually exclusive periods:

- a. **Induction** period: From day of first dose of midostaurin to the day before start of consolidation period (i.e. end of induction phase plus any rest/recovery days). Up to 2 cycles (28 days of treatment/cycle and a recovery period)
- b. **Consolidation** period: From day of first dose of study treatment in consolidation phase to the day before start of maintenance (i.e. end of consolidation phase plus any rest/recovery days).
  - Up to 4 cycles (28 days of treatment/cycle and a recovery period)
- c. **Maintenance** period: From day of first dose of midostaurin in the maintenance phase to the date of last dose of midostaurin + 30 days.

Up to 12 cycles (28 days of treatment/cycle)

It is noted that if a patient permanently discontinues study treatment during any of these periods, on-treatment is considered until the date of last dose of study treatment + 30 days (unless patient withdraws study informed consent or dies before then, then it is till the withdrawal/death date)

3. **Post-treatment**: from last date of study treatment + 31 days to end of study Each period will contain all patients who entered that period (incl. withdrawal, drop-outs etc.)

## Study drug and study treatment

Study drug refers to the individual drugs used in the study after signing of informed consent, i.e. the Novartis investigational drug midostaurin, or its partners, cytarabine and daunorubicin (or idarubicin).

Study treatment refers to any component of the study drugs, midostaurin, cytarabine and daunorubicin (or idarubicin).

## Date of first administration of study drug

The date of first administration of study drug is derived as the first date when a nonzero dose of study drug is administered. The date of first administration of study drug is also referred to as *start date of study drug*. Start date of study drug is defined for each drug which is part of study treatment, by period (induction, consolidation, maintenance, where applicable) and overall.

## Date of last administration of study drug

The date of last administration of study drug is defined as the last date when a nonzero dose of study drug is administered. This date is also referred to as *last date of study drug*. Last date of study drug is defined for each drug which is part of study treatment, by period (induction, consolidation, maintenance, where applicable) and overall.

## Date of first administration of study treatment

The date of first administration of study treatment (will be midostaurin for all patients) is derived as the first date when a nonzero dose of any component of study treatment is administered. It is derived by period (induction, consolidation, maintenance) and overall.

For example, if the 1<sup>st</sup> dose of midostaurin is taken on 08-Feb-2016, and 1<sup>st</sup> dose of a combination partner (e.g. cytarabine), is taken on 01-Feb-2016, then the date of first administration of study treatment is 01-Feb-2016. The date of first administration of study treatment is also referred to as *start date of study treatment*.

## Date of last administration of study treatment

The date of last administration of study treatment is derived as the last date when a nonzero dose of any component of study treatment is administered. It is derived by period (induction, consolidation, maintenance) and overall.

For example if the last dose of midostaurin is taken on 21-Mar-2016, and the last dose of a combination partner is taken on 03-Apr-2016, then the date of last administration of study treatment is on 03-Apr-2016. This date is also referred to as *last date of study treatment*.

## **Duration of exposure**

## Daunorobucin, Idarubicin and Cytarabine

The duration of exposure for the **study drugs** will be calculated by cycle, period (induction, consolidation, maintenance, when applicable) and overall as:

- Duration of study drug exposure (days) in a **cycle** = [(date of last administration of study drug in that cycle) (date of first administration of study drug in that cycle) + 1]
- Duration of study drug exposure (days) in a **period** = sum of durations of study drug exposure (days) in each cycle of that period
- Overall duration of study drug exposure (days) = sum of durations of study drug exposure (days) in each cycle

## **Study treament and Midostaurin**

The duration of exposure for the **study treatment and Midostaurin** will be calculated by cycle, period (induction, consolidation, maintenance) and overall as:

- Duration of study treatment/Midostaurin exposure (days) in a **cycle** = [(date of last administration of study treatment/Midostaurin in that cycle) (date of first administration of study treatment/Midostaurin in that cycle) + 1]
- Duration of study treatment exposure (days) in a **period** = sum of durations of study trt/Mido exposure (days) in each cycle of that period.
- Overall duration of study treatment exposure (days) = [(date of last administration of study treatment/Midostaurin) (date of first administration of study treatment/Midostaurin) + 1]
- If the start or end date of a study drug is missing, the duration will be missing. The durations will include periods of temporary interruption (planned or actual) for any reason.

## **Dose interruption**

For **midostaurin**: An interruption is defined as a zero dose on one or more days between two non-zero dosing records. Any rest period as part of the regimen/schedule is not considered as an interruption e.g. Days 1 to 7 at the start of a cycle in the induction and consolidation phases is not considered as an interruption.

For **daunorubicin** (or **idarubicin**) and **cytarabine**: An interruption is defined as a zero dose administered on one or more scheduled days of administration e.g. a zero dose on Days 1, 3 or 5 for cytarabine in the consolidation phase.

Note: The last zero dose of a study drug (followed by permanent discontinuation) is not considered as a dose interruption. Additionally, two consecutive zero doses will be counted as one interruption if the reasons for these two consecutive dose interruptions are the same.

For the purpose of summarizing interruptions and reasons, in case multiple entries for interruption are entered on consecutive days with different reasons these will be counted as separate interruptions. However, if the reason is the same in these multiple entries on consecutive days, then it will be counted as one interruption.

#### **Dose reduction**

A dose reduction is where the prescribed dose is lower than the previous prescribed dose or where the actual dose administered/total daily dose is lower than the prescribed dose. Any dose change to correct a dosing error will not be considered a dose reduction, e.g. if due to a dosing error, a patient receives higher than protocol planned starting dose and moves down to the planned starting dose then this is not counted as a reduction, however if they move directly from a higher than planned starting dose down to a lower than protocol planned starting dose, then this is counted as a reduction.

Note: It is assumed that if there is a dose reduction, then the 'Dose changed' box was ticked on the dose administration electronic case report form (eCRF) page.

If dose is recorded by regimen is missing or entered as 'none', it is assumed that the study drug was taken as per-protocol.

#### **Actual cumulative dose**

Cumulative doses will be derived for each of the study drugs: midostaurin, daunorubicin and idarubicin.

The actual cumulative dose refers to the total actual dose administered, over the duration for which the patient is on study drug as documented in the dose administration eCRF.

For patients who did not take any study drug, the actual cumulative dose is by definition equal to zero.

The actual cumulative dose is the sum of the non-zero doses recorded over the study drug dosing periods. Rest periods are not included.

## **Actual dose intensity (DI)**

Dose intensity (DI) will be derived for each of the study drugs: midostaurin, daunorubicin and idarubicin.

DI for patients with non-zero duration of exposure is defined as follows:

DI (*dosing unit / unit of time*) = Actual cumulative dose (*dosing unit*) / Duration of exposure (*unit of time*).

```
For example, DI (mg/day) = Actual cumulative dose (mg) / Duration of exposure (day) = 1300 mg / 14 days = 92.9 mg/day
```

For patients who did not take any study drug the DI is by definition equal to zero.

### Study day

The study day describes the relative day of the event related to the start date of midostaurin.

The reference start date is designated as **Study Day 1.** Study Day –1 is the day that precedes Day 1. Study Day 0 is not defined. Study day is not to be used in numerical computations, for example in calculating exposure.

The study day will be calculated as:

- The date of the event (visit date, onset date of an event, assessment date etc.) reference start date + 1, if event is on or after the reference start date
- The date of the event (visit date, onset date of an event, assessment date etc.) reference start date, if event precedes the reference start date

The reference start date for all assessments (adverse events (AEs), laboratory etc.) will be the start date of study treatment.

The study day will be displayed in the data listings. If an event starts before the reference start date, the study day displayed in the listing will be negative.

#### 2.1.2 Baseline

Baseline is the result of an investigation describing the "true" uninfluenced state of the patient, defined as the period from the date of signing any informed consent document to the start date of midostaurin.

The last non-missing assessment, including unscheduled assessments on or before the first dose of midostaurin is defined as "baseline value" or "baseline assessment". Assessments, specified to be collected post-dose on the first date of midostaurin are not considered for baseline.

Where electrocardiogram (ECG) replicates are provided, the average of the ECG parameters at that assessment will be used in the analyses.

If patients have no value as defined above, the baseline value will be missing.

#### 2.1.3 On-treatment assessment/event

The definition of on-treatment is given below, depending on the context.

For safety summary tables (over the entire duration of the study) an on-treatment AE is defined as any AE reported in the following time interval (including the lower and upper limits):

<date of first administration of midostaurin; date of last administration of study treatment</li>
 + 30 days>

This corresponds to the definition of treatment-emergent AEs given in the protocol, i.e. AEs which are newly reported or worsening from baseline.

An on-treatment assessment is defined as any assessment performed after the date of first administration of midostaurin (except for assessments specified to be collected post-dose on that day), i.e. assessments performed in the following time interval (including the lower and upper limits):

• <date of first administration of midostaurin + 1; date of last administration of study treatment + 30 days>

For patients whose last date of study treatment is missing, on-treatment assessments/events include any assessment/event present in the database occurring after the start date of study treatment.

Listings will contain all data, flagging assessments/events outside of the on-treatment period where applicable.

## 2.1.4 Definition of months and years

A month will be calculated as (365.25 / 12) = 30.4375 days. If duration is to be reported in months, duration in days will be divided by 30.4375. If duration is to be reported in years, duration in days will be divided by 365.25.

#### 2.1.5 Time windows

Time windows for assessments are based on protocol specified windows, see protocol Table 7-1.

If more than one assessment is done within the same time window, the assessment performed closest to the target date will be used. For two assessments within a time window are equidistant from the target date then the earlier of the two assessments will be used. If there are multiple assessments for the same date, then the worst case will be used.

For unplanned visits, will be classified as follows:

| Assessment | Target day of assessment | Time Interval |
|---|---|---|
| Baseline | Date when visit = IND C1D8 (or | Last date <= date of IND C1D8 |
| | Day1) | |
| INDC1 | Date when visit = INDC1D8 | Date of IND C1D8 - 7 <= date < date of |
| | | IND C2D1 |
| INDC2 | Date when visit = INDC2D8 | Date of IND C2D1 <= date < date of CON |
| | | C1D1 |
| CONC1 | Date when visit = CONC1D8 | Date of CON C1D1 <= date < date of |
| | | CON C2D1 |
| CONC2 | Date when visit = CONC2D8 | Date of CON C2D1 <= date < date of |
| | | CON C3D1 |
| CONC3 | Date when visit = CONC3D8 | Date of CON C3D1 <= date < date of |
| | | CON C4D1 |
| CONC4 | Date when visit = CONC4D8 | Date of CON C4D1 <= date < date of |
| | | MAIN C1D1 |
| MAINC1 | Date when visit = MAIN C1D1 | Date of MAIN C1D1 <= date < date of |
| | | MAIN C2D1 |

| | ••• | |
|---|---|---|
| MAINC12 | Date when visit = MAIN C12D1 | Date of MAIN C12D1 <= date <= date of |
| | | last non-zero dose +30 |
| End Of | Date when visitnum =399 | Date when visitnum in (399, |
| Treatment | | 399.001,399.002,) |

## 2.1.6 Definition of end of study

The study will end around 18 to 25 months (mo) after LPFV depending on number of cycles and recovery durations (2mo induction + 2mo recovery + 4mo consolidation + 4mo recovery + 12mo maintenance + 1mo safety follow-up). Study treatment will be provided until disease progression, death, unacceptable toxicities, physician's decision, patient/guardian's decision, protocol deviation, study termination by sponsor, lost to follow-up, technical problems, pregnancy, patient withdrew consent or until the end of study, whichever event occurs first. All patients must have safety follow-up for 30 days, after the last dose of study treatment except if study consent was withdrawn.

## 2.1.7 Early study termination

The study can be terminated at any time for any reason by Novartis. Should this be necessary, the patient should be seen as soon as possible and the same assessments should be performed as for a discontinued or withdrawn patient.

## 2.1.8 Chemotherapy group assignment

Patients will be assigned to '7+3' or '5+2' chemotherapy groups considering the following rules of the first induction cycle:

- If cytarabine duration is ≥ 7 days, '7+3' group will be assigned, without considering the duration of daunorubicin/idarubicin.
- If cytarabine duration is < 7 days, '5+2' group will be assigned, without considering the duration of daunorubicin/idarubicin.

## 2.2 Analysis sets

## 2.2.1 All enrolled patients

The 'All enrolled patients' set comprises all screened patients who are not screening failures.

## 2.2.2 Full analysis set

The Full Analysis Set (FAS) comprises all patients who received at least one dose of midostaurin and have a documented FLT3 mutation (ITD or TKD).

## 2.2.3 Safety set

The safety set comprises all patients who received at least one dose of midostaurin.

## Screening failures

Patients who sign an informed consent form but fail to start on midostaurin for any reason.

## 2.3 Subgroup analysis

Safety and efficacy data will be reported for the following subgroups:

- Age [(i)  $\leq$  60 / > 60 years old and/or (ii)  $\leq$  60 / > 60 to  $\leq$  70 / > 70 years old]
- Gender (female / male)
- Chemotherapy groups ('7+3' / '5+2')
- Type of induction drugs (Daunorubicin (<60 mg/m²), daunorubicin (>= 60 mg/m²) and Idarubicin)

# 2.4 Patient disposition, demographics and other baseline characteristics

## 2.4.1 Patient disposition

Disposition data will be listed and summarized descriptively by screening and period (induction, consolidation and maintenance) for the FAS.

Summaries will also include the number of patients who did not receive any dose of study treatment, having received at least one dose of study treatment, treatment completed as per protocol criteria or treatment permanently discontinued with reason, as reported in the dose administration record eCRF pages.

Informed consent and inclusion/exclusion criteria data will be listed. Screening data for screen failure patients will be listed.

## 2.4.2 Patient demographics and other baseline characteristics

Demographic and other baseline data (e.g. medical history, diagnosis and extent of cancer, eastern cooperative oncology group (ECOG) performance status, FLT3 mutation status etc.) will be summarized descriptively or listed as appropriate for the FAS.

Age will also be categorized as:

- <=60, > 60 years and/or
- <= 60 / >60 to <= 70 / > 70 years old.

Demographic data for screen failure patients will also be listed.

# 2.5 Treatments (study treatment, concomitant therapies, compliance)

## 2.5.1 Dosing regimen

All patients on study will receive standard chemotherapy plus midostaurin.

The protocol treatment allows 1-2 cycles of standard induction therapy with cytarabine and daunorubicin (or idarubicin) and up to 4 cycles of cytarabine consolidation, with midostaurin

given sequentially during each cycle, and up to 12 cycles of maintenance therapy with single-agent midostaurin as given in Figure 1-1.

Table 2-1 Dose and treatment schedule – Induction

| Treatment | Dose, route and frequency (based on 28-day cycles) |
|---|---|
| Cytarabine (Ara-C) with anthracycline (Idarubicin or Daunorubicin) (7+3) | Ara-C:100-200 mg/m²/day by CIVI days 1-7 (168 hour infusion) Daunorubicin: 60-90 mg/m²/day by IV push on days 1-3 or Idarubicin: 12 mg/m²/day by IV push on days 1-3 |
| Cytarabine with<br>anthracycline (Idarubicin or<br>Daunorubicin) (5+2) | Ara-C:100 mg/m²/day by CIVI days 1-5 Daunorubicin: 60 mg/m²/day by IV push on days 1-2 or Idarubicin: 12 mg/m²/day by IV push on days 1-2 |
| Midostaurin | 50 mg (two 25 mg capsules) twice a day by mouth on days 8-28 |

Table 2-2 Dose and treatment schedule – Consolidation

| Treatment Dose, route and frequency (based on 28-day cycles) | |
|---|---|
| Cytarabine | 1-3 g/m $^2$ every 12 h on days 1, 3, 5 x up to 4 cycles based on age and per investigator discretion |
| Midostaurin | 50 mg (two 25 mg capsules) twice a day by mouth on days 8-28 |

Table 2-3 Dose and treatment schedule – Maintenance

| Treatment | Dose, route and frequency (based on 28-day cycles) |
|---|---|
| Midostaurin | 50 mg (two 25 mg capsules) twice a day by mouth on days 1-28 |

## 2.5.2 Study treatment and tolerability

## Study treatment

Duration of exposure (days), actual cumulative dose and actual dose intensity will be summarized by period and overall for each of the study drugs: midostaurin, daunorubicin and idarubicin for the safety set. Duration of exposure (days), actual cumulative dose and actual dose intensity will be summarized also by cycle. The number of patients with midostaurin dose changes, interruptions and permanent discontinuations will be presented by age category and overall, along with reasons for the dose change/interruption/permanent discontinuation.

Duration of midostaurin treatment exposure (days) will also be categorized and summarized by period and overall for the safety set using the following intervals:

• <20; >20; >40; >60; >120; >180; >240; >300; >360

Duration of study treatment exposure (days) will be summarized by period and overall for the safety set using the following intervals:

•  $\leq 28$ ;  $\geq 28$ ;  $\geq 56$ ;  $\geq 84$ ;  $\geq 112$ ;  $\geq 196$ ;  $\geq 280$ ;  $\geq 364$ ;  $\geq 448$ ;  $\geq 532$ 

Duration include the rest/recovery days between cycles and will be derived as the following:

Last intake of any study treatment component – first intake of any study treatment component +1

If there are more than 10 patients in each regimen exposure will be further summarized by regimen ("7+3" and "5+2").

Data will be listed for all patients in the safety set.

### **Tolerability**

Tolerability of midostaurin will be evaluated in terms of dose reductions or dose interruptions due to an AE.

## 2.5.3 Prior, concomitant and post therapies

Medications and significant non-drug therapies prior to and after the start of the study treatment will be coded according to the world health organization (WHO) Drug Reference List and summarized by anatomical therapeutic chemical (ATC) classification and preferred term.

A summary table and listing for prior antineoplastic therapies will be provided for the full analysis set.

Summary tables for concomitant medications and concomitant non-drug therapies by treatment period and overall for the full analysis set will be provided. Prior, concomitant and post study treatment medications and non-drug therapies will be listed for the safety set. Records outside of on-treatment period will be flagged.

#### 2.5.4 Protocol deviations

Protocol deviations will be listed for all screened patients. In addition, the number (%) of protocol deviations with COVID-19 relationship will be presented by type of deviation for all enrolled subjects.

## 2.6 Analysis of the primary objective

## 2.6.1 Primary endpoint

The analysis of the primary endpoint is described in Section 2.8.

## 2.6.2 Statistical hypothesis, model, and method of analysis

Not applicable.

## 2.6.3 Handling of missing values/censoring/discontinuations

See Section 2.8.

## 2.6.4 Supportive analyses

Not applicable.

## 2.7 Analysis of the secondary objectives

## 2.7.1 Secondary endpoints

The secondary objectives in this study are to assess the clinical efficacy of midostaurin in combination with chemotherapy regimens in induction and consolidation and the clinical efficacy of midostaurin in maintenance phase.

Clinical efficacy rate will be presented for the FAS. All assessments before the last available on-treatment assessment will be included. Listings will include all data and will be based on the FAS. Records outside of on-treatment period will be flagged. For patients who discontinued prior to the first efficacy assessment, the response will be reported as 'unknown'.

Clinical efficacy rate is defined as the proportion of patients with complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) as per local review. The CR and CRi are defined by the national comprehensive cancer network (NCCN) guidelines version 1.2017 for AML.

Clinical efficacy rate and its 95% confidence interval will be presented by period (induction, consolidation and maintenance) and overall as described in Section 2.1.1. The best overall response will be analyzed in each period and overall. If there are more than 10 patients in each regimen and age category, the clinical efficacy rate will be further summarized by regimen ("7+3" and "5+2") and age category (e.g. <=60, >60 years and/or <=60 / >60 to <=70 / >70 years old) and by sex.

## 2.7.2 Statistical hypothesis, model, and method of analysis

Not applicable.

## 2.7.3 Handling of missing values/censoring/discontinuations

Not applicable.

## 2.8 Analysis of secondary efficacy objective(s)

Not applicable.

## 2.9 Safety analyses

The primary objective is to further assess the safety of midostaurin in induction, consolidation and maintenance therapy including the '7+3' regimen, daunorubicin (60-90mg/m²/day), the substitution of daunorubicin by idarubicin (12 mg/m²/day) and cytarabine (100-200 mg/m²/day) and also allowing the "5+2" reduced dose regimen.

Except for baseline values, safety summary tables will only include on-treatment assessments (up to 30 days after study treatment discontinuation) and will be based on the safety set. Listings will include all data and will be based on the safety set.

#### 2.9.1 Adverse events (AEs)

The AEs will be re-coded using the latest version of the medical dictionary for regulatory activities (MedDRA) at the time of the analysis.

AEs will be graded using the common toxicity criteria for adverse events (CTCAE) Version 4.03. AEs will be summarized by period and overall for the safety set. AEs tables will be provided by age category. AEs with different starts dates in different periods will be counted within each period. If a patient reported more than one AE with the same preferred term (PT), the AE with the greatest severity will be presented. If a patient reported more than one AE within the same primary system organ class (SOC), the patient will be counted only once with the greatest severity at the SOC level, where applicable. An AE with missing CTCAE grade will be included in the 'All grades' column of the summary tables.

In AE summaries, the primary SOC will be presented alphabetically and the PTs will be sorted within the primary SOC in descending frequency.

Summary tables will be provided for:

- Overview of AEs and age category
  - In-text table
- All AEs regardless of relationship to study treatment by primary system organ class (SOC), preferred term (PT) and maximum severity and age category
  - In-text table by SOC and maximum severity
  - In-text table by PT and maximum severity
- AEs suspected to be related to study treatment by SOC, PT and maximum severity and age category
  - In-text table by PT and maximum severity
- AEs leading to treatment discontinuation regardless of relationship to study treatment by SOC, PT and maximum severity and age category
  - In-text table by PT and maximum severity
- AEs leading to treatment reduction or interruption regardless of relationship to study treatment by SOC, PT and maximum severity and age category
  - In-text table by PT and maximum severity
- Serious AEs (SAEs) regardless of relationship to study treatment by SOC, PT and maximum severity and age category
  - In-text table by PT and maximum severity
- On-treatment deaths by SOC and PT and age category
  - In-text table by SOC and PT
- All deaths by SOC, PT and age category
- \*Non-SAEs regardless of relationship to study treatment (threshold=5%) by SOC and PT
- \*On treatment deaths and SAEs by SOC and PT

\*(For the legal requirements of ClinicalTrials.gov and EudraCT, two required tables on <ontreatment/treatment emergent> AEs which are not SAEs with an incidence greater than 5% and on <on-treatment/treatment emergent> SAEs and SAE suspected to be related to study treatment will be provided by SOC and PT on the safety set.

If for a same patient, several consecutive AEs (irrespective of study treatment causality, seriousness and severity) occurred with the same SOC and PT:

- a single occurrence will be counted if there is  $\leq 1$  day gap between the end date of the preceding AE and the start date of the consecutive AE
- more than one occurrence will be counted if there is > 1 day gap between the end date of the preceding AE and the start date of the consecutive AE

For occurrence, the presence of at least one SAE/SAE suspected to be related to study treatment/non SAE has to be checked in a block e.g., among AEs in a  $\leq$  1 day gap block, if at least one SAE is occurring, then one occurrence is calculated for that SAE.

The number of deaths resulting from SAEs suspected to be related to study treatment and SAEs irrespective of study treatment relationship will be provided by SOC and PT.

Listings will be provided for all AEs, SAEs and AEs leading to discontinuations (including those from the pre and post-treatment periods). Records outside of on-treatment period will be flagged.

#### Adverse events of special interest / grouping of AEs 2.9.1.1

The adverse events of special interest (AESI) are maintained and updated on a regular basis in the project case retrieval sheet (CRS) and the latest version at the time of the analyses will be used. The CRS to produce AESI outputs will be stated in listing 14.3.2-8.

A summary table for AESIs will be provided by period and overall for the safety set.

#### 2.9.2 **Deaths**

See Section 2.8.1. A listing will be provided of all deaths. Deaths outside of the on-treatment period will be flagged.

#### 2.9.3 Laboratory data

Laboratory values are converted to the international system of units (SI). CTCAE Grade 0 will be assigned for all non-missing values not graded as 1 or higher. Grade 5 will not be used. For laboratory results where grades are not defined by CTCAE v4.03, results will be categorized as low/normal/high based on laboratory normal ranges.

The following summaries will be generated separately for key hematology and biochemistry by period and overall for the safety set:

- Shift tables by grade (or low/normal/high if grades not available) to compare baseline to the worst on-treatment value:
  - Hematology: Neutrophils (absolute) and platelets
  - Chemistry: Creatinine, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase

Listing of all laboratory data (including urinalysis, coagulation, thyroid panel, pregnancy test etc.) will be provided with the corresponding CTCAE grades, if applicable, and the classifications relative to the laboratory normal ranges. Records outside of on-treatment period will be flagged.

## 2.9.4 Other safety data

## 2.9.4.1 Electrocardiogram (ECG)

Electrocardiogram (ECG) data will be listed. Listing will include date of assessment, position=supine, any new clinically significant abnormalities (yes/no), QTcF (Fridericia's correction), mean heart rate and mean PR, QT and QRS durations. Notable values and records outside of on-treatment period will be flagged.

Where ECG replicates are provided for an assessment, the average of the ECG parameters at that assessment will be used in the analyses.

Table 2-4 Notable criteria for ECG parameters<sup>1</sup>

| Parameter | Notable low value | Notable high value |
|---|---|---|
| | | New value of >450 and ≤ 480 ms |
| | | New value of >480 and ≤ 500 ms |
| QTcF | | New value of >500 ms |
| | | Increase from baseline of >30 ms to ≤ 60 ms |
| | | Increase from baseline of >60 ms |
| Heart rate | Decrease >25% from baseline and to a value <50 bpm | Increase >25% from baseline and to a value >100 bpm |
| PR | | Increase >25% from baseline and to a value >200 ms New value of >200 ms |
| QRS | | Increase >25% from baseline and to a value >120 ms New value of >120 ms |

## 2.9.4.2 Cardiac imaging

The left ventricular ejection fraction (LVEF) data will be summarized for change from baseline to the worst on-treatment value by period and overall for the safety set. A listing will be provided showing the imaging method (multi gated acquisition scan (MUGA) or echocardiogram), date of assessment, LVEF percentage, the overall interpretation (normal, clinically insignificant abnormality or clinically significant abnormality) and the corresponding ejection fraction CTCAE v4.03 grades. Records outside of on-treatment period will be flagged.

#### Grades:

- Grade 0: Non missing value below Grade 2
- Grade 1: NA
- Grade 2: 50-40% or 10-19% drop from baseline i.e.
  - $40\% \le LVEF \le 50\%$  or -20% < absolute change from baseline  $\le -10\%$
- Grade 3: 39-20% or  $\geq$ 20% drop from baseline i.e.
  - $20\% \le LVEF < 40\%$  or absolute change from baseline  $\le -20\%$
- Grade 4: <20% i.e.
  - LVEF < 20%

## 2.9.4.3 Chest X-ray

Chest x-ray data will be listed showing date of assessment and the overall interpretation (normal, clinically insignificant abnormality or clinically significant abnormality). Records outside of on-treatment period will be flagged.

## 2.9.4.4 **Vital signs**

Vital signs (height, weight, body surface area, temperature, position, pulse and systolic/diastolic blood pressure) will be summarized by period and overall for the safety set. Listings will be provided with notable values and records outside of on-treatment period flagged.

Table 2-5 Notable criteria for vital signs<sup>1</sup>

| Vital sign (unit) | Notable low value | Notable high value |
|---|---|---|
| Weight (kg) | decrease ≥ 10% from baseline | increase ≥ 10% from baseline |
| Body temperature (°C) | | ≥ 39.1 |
| Pulse rate (bpm) | ≤ 50 and decrease from baseline of >25% | ≥ 100 and increase from baseline of >25% |
| Systolic blood pressure (mmHg) | ≤ 90 and decrease from baseline of ≥ 20 | ≥ 180 and increase from baseline of ≥ 20 |
| Diastolic blood pressure (mmHg) | ≤ 50 and<br>decrease from baseline of ≥ 15 | ≥ 105 and increase from baseline of ≥ 15 |

## 2.9.4.5 ECOG performance status

ECOG performance status data will be listed. Records outside of on-treatment period will be flagged. Baseline summary will be provided as part of the demographics table.

Table 2-6 ECOG Performance Status

| Grade | ECOG |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

## 2.10 Pharmacokinetic endpoints

Not applicable.

## 2.11 PD and PK/PD analyses

| * T . | | 1. 11 | |
|-------|-----|---------|---|
| Not | ann | licable | |
| 1101 | upp | ncacic | • |

# 2.13 Biomarkers

Not applicable.

## 2.14 Other Exploratory analyses

| resource utilization will be used to evaluate the symptom burden, overall quality of life and change in status of a patient's overall so with. | |
|---|---|
| The safety set will be used for analyzing utilization data unless otherwise specified. | resource |



#### 2.14.3 Resource utilization

Descriptive statistics will be used to summarize resource utilization, e.g. the reason for hospitalization due to AE or not, if number of hospital days by facility/ward type and discharge status used during hospital stay(s). Listings will flag records outside of the on-treatment period.

## 2.15 Interim analysis

No formal interim analysis is planned for this study. Analyses may be performed periodically (e.g. annually), if needed, to fulfill regulatory requests, safety updates or for publication purposes.

## 3 Sample size calculation

Approximately 300 patients will be enrolled in this study. The planned sample size is based on the average expected accrual rate (17 patients per month) and the planned recruitment duration (18 months) of the trial. The actual sample size may differ from this planned number. A sample size of 300 patients provides a 95% probability of observing at least one patient with an adverse event (AE) assuming a true probability of occurrence of 1%.

Table 3-1 provides probabilities to detect at least one patient with an AE for different sample sizes and different true AE incidences.

Table 3-1 Probability to detect at least one patient with an AE for different sample sizes and different true AE incidences

| Incidence of an | Sample size | | |
|-----------------|-------------|--------|--------|
| adverse event | N=200 | N=250 | N=300 |
| 0.4% | 0.5514 | 0.6329 | 0.6995 |
| 0.5% | 0.6330 | 0.7144 | 0.7777 |
| 0.6% | 0.6999 | 0.7779 | 0.8356 |
| 0.8% | 0.7994 | 0.8657 | 0.9102 |
| 1.0 % | 0.8660 | 0.9189 | 0.9510 |
| 1.3% | 0.9270 | 0.9620 | 0.9803 |

## 4 Change to protocol specified analyses

None.

## 5 References

- 1. Oncology guideline for safety analysis, v1.0, dated 09-Jun-2016
- 2. Oncology standard outputs TFL v3.1, dated 03-Aug-2017
- 3. NCCN Clinical Practice Guidelines in Oncology: Acute Myeloid Leukemia. Version 1.2017, https://www.nccn.org/professionals/physician\_gls/pdf/aml.pdf, last accessed on 27 March 2017
- 4. Cheson et al. (2003) Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Journal of Clinical Oncology 21:24, 4642-4649

## 6 Appendix

## 6.1 Imputation rules

## 6.1.1 AE, CM date imputation

Table 6-1 Imputation of start dates (AE, CM)

| Missing<br>Element | Rule |
|---|---|
| day, month,<br>and year | No imputation will be done for completely missing dates |
| day, month | <ul> <li>If available year = year of study treatment start date then <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 01JanYYYY</li> <li>Else set start date = study treatment start date.</li> </ul> </li> <li>If available year &gt; year of study treatment start date then 01JanYYYY</li> <li>If available year &lt; year of study treatment start date then 01JulYYYY</li> </ul> |
| day | <ul> <li>If available month and year = month and year of study treatment start date then <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 01MONYYYY.</li> <li>Else set start date = study treatment start date.</li> </ul> </li> <li>If available month and year &gt; month and year of study treatment start date then 01MONYYYY</li> <li>If available month and year &lt; month year of study treatment start date then 15MONYYYY</li> </ul> |

Table 6-2 Imputation of end dates (AE, CM)

| Missing | Rule |
|---|---|
| Element | (*=last treatment date plus 30 days not > (death date, cut-off date, |
| | withdrawal of consent date)) |
| day, month, and year | • Completely missing end dates (incl. ongoing events) will be imputed by the end date of the on-treatment period* |
| day, month | • If partial end date contains year only, set end date = earliest of 31DecYYYY or end date of the on-treatment period * |
| day | • If partial end date contains month and year, set end date = earliest of last day of the month or end date of the on-treatment period* |

In the case of the imputed end date is before than start date, then the end date will be imputed equals to start date.

Any AEs and ConMeds with partial/missing dates will be displayed as such in the data listings.

Any AEs and ConMeds which are continuing as per data cut-off will be shown as 'ongoing' rather than an imputed end date provided.

## 6.1.2 Prior therapies date imputation

Missing day is defaulted to the 15<sup>th</sup> of the month and missing month and day is defaulted to 01-Jan for start and end dates in ZT domain.

## 6.2 Laboratory parameters derivations

CTC grading for blood differentials is based on absolute values. However, this data may not be reported as absolute counts but rather as percentage of WBC.

If laboratory values are provided as '<X' (i.e. below limit of detection) or '>X', prior to conversion of laboratory values to SI unit, these numeric values are set to X.

The following rules will be applied to derive the WBC differential counts when only percentages are available for a xxx differential

```
xxx count = (WBC count) * (xxx %value / 100)
```

Further derivation of laboratory parameters might be required for CTCAE grading. For instance, corrected calcium can be derived using the reported total calcium value and albumin at the same assessment using the following formula:

Corrected Calcium (mg/dL) = Calcium (mg/dL) - 0.8 [Albumin (g/dL)-4]

In order to apply the above formula, albumin values in g/L will be converted to g/dL by multiplying by 0.1, calcium values in mmol/L will be converted to mg/dL by dividing by 0.2495. For calculation of laboratory CTC grades 0 and 1, the normal range for derived corrected calcium is set to the same limits (in mg/dL) as for calcium.

For missing Blood Urea Nitrogen (BUN) or urea values the following formulae will be applied:

Urea (mg/dL) = BUN (mg/dL) / 0.357

BUN (mg/dL) = Urea (mg/dL) / 2.1428



